CLINICAL TRIAL: NCT02447341
Title: Multicenter Observational Study to Determine the Profile and Antithrombotic Management of Patients With Nonvalvular Atrial Fibrillation Attending Internal Medicine Departments in Spanish Hospitals (Perfilar Study)
Brief Title: Profile and Antithrombotic Management of Patients With NVAF Attending Internal Medicine Departments in Spain (PERFILAR Study)
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-372
Record Dates: First submitted 2015-05-05; First posted 2015-05-18 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Anticoagulation, Blood Thinners , Atrial Fibrillation, Bleeding, Stroke
MeSH Terms: conditions — Atrial Fibrillation; Hemorrhage; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- In patients
- Out patients

SUMMARY:
This is a national, multicenter, cross-sectional, observational study within a convenience sample of Internal Medicine departments from 100 hospitals in Spain which agree to participate in the study. This study will be a cross-sectional chart review which will require the collection of data from medical records and from face-to-face interviews conducted during the inclusion visit. Physician interviews are needed to collect three variables of interest, recommended by the Spanish Society of Internal Medicine as necessary data about profile and management of NVAF patients: cognitive deterioration based on the patient's responses, physician's assessment of the patient's life expectancy, and physician's opinion of the antithrombotic treatment previously prescribed. The investigators will only provide their opinion on previously prescribed therapies (i.e. prescribed before F2F). Hospitals to be contacted for the study include those known to participate in observational studies in Spain; the hospitals will therefore not be a random sample of Spanish hospitals.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Adult patients (≥18 years old)
* Patients diagnosed with Non-valvular atrial fibrillation (NVAF) any time prior to the inclusion date (prevalent or incident patients)
* Patients treated or not treated with an antithrombotic therapy
* Treated patients should have begun treatment prior to the inclusion visit
* Patients attending Internal Medicine departments, either for a hospital appointment (outpatients) or hospitalization (inpatients) for any reason)
* Patients which signed the informed consent

Exclusion Criteria:

* Patients diagnosed with valvular atrial fibrillation any time in their medical records
* Patients with anticoagulant treatment prescribed for venous thromboembolic disease any time prior to the inclusion date
* Patients which participated in any clinical trial with anticoagulant and/or antiplatelet agents in the previous six months
* Patients incapable of giving their informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with NVAF
Sampling Method: Non-Probability Sample
Enrollment: 987 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Demographics (age, sex, living environment) of patients with NVAF attending Spanish hospitals by antithrombotic treatment type (including absence of treatment) | Approximately 6 months
Clinical characteristics (bleeding, myocardial infarction, stroke) of patients with NVAF attending Spanish hospitals by antithrombotic treatment type (including absence of treatment) | Approximately 6 months

SECONDARY OUTCOMES:
Clinical Characteristics (bleeding, myocardial infarction, stroke) associated with the administration of oral antithrombotic treatments | Approximately 6 months
  Clinical Characteristics (bleeding, myocardial infarction, stroke) associated with the administration of oral antithrombotic treatments (i.e.Vitamin K Antagonists (VKAs), New Oral Anticoagulants (NOACs), antiplatelet drugs, or combinations of anticoagulant and antiplatelet drugs
Estimating the rate of compliance to treatment and by calculating the proportion of patients treated in accordance with guidelines among the patients treated with oral anticoagulants | Approximately 6 months
  Evaluate current clinical practice in Internal Medicine departments in Spanish hospitals according to the European Guidelines by estimating the rate of compliance to treatment; and by calculating the proportion of patients treated in accordance with guidelines among the patients treated with oral anticoagulants

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Barcelona, Spain

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx